CLINICAL TRIAL: NCT00137488
Title: Angiogenic Profile and Non-invasive Imaging May Predict Tumor Progression of High Risk Group Low Grade Glioma (LGG)
Status: Completed | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: CNS-09-0024/ethics 21656
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2012-04

CONDITIONS: Glioma
Keywords: non-enhancing lesion; low grade glioma; high risk group selection
MeSH Terms: conditions — Glioma | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: imaging and angiogenic profiles — Image tumor angiogenesis by DCE-MRI using 1.5- or 3-T MRI instruments (13,14,15) pre-and postoperatively (before biopsy or surgery).

SUMMARY:
The low grade glioma (LGG) is a type of brain tumor which is generally more common in younger age group patients. Most patients with LGG undergo surgery which is mostly incomplete due to concern about loss of function. This is an incurable disease. More than half of these patients progress to a higher grade with a worse outcome within five years of their diagnosis and only one-third survive for up to ten years. Post-operative radiation treatment improves local control without survival advantage. Efforts are being made without great success to select the patients with a higher risk of progression based on physical characteristics and histological features.

Tumor vascularity is thought to be the key element in tumor progression. Tremendous progress has been made in functional imaging by using magnetic resonance imaging (MRI) 3-Tesla (3T) and in biotechnology which can be used to investigate angiogenic gene profiles in order to identify gene signature for these tumors. In this study the investigators are proposing that patients of LGG with a higher risk of tumor progression may be selected by functional imaging and angiogenic profiles. These higher risk patients may be candidates for post-operative radiation in the future with a potential survival benefit.

DETAILED DESCRIPTION:
Summary: Comprehensive analysis of the angiogenesis-related gene expression profiles and tumor perfusion of patients with LGG will provide a novel understanding of subgroup (low and high-risk) of LGG. Thus, this study will allow identifying clinically relevant factors predictive for tumor progression and to select patients in high-risk group for adjuvant radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age
* Brain tumor with no contrast enhancement on conventional MRI and confirmed histological of LGG
* No adjustment treatment
* Consent to participate in study
* No contra-indication for dynamic contrast-enhanced (DCE)-MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients referred to Cross Cancer Institute between 2004 and 2005
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2005-11; Primary Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bassam Abdulkarim, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada